CLINICAL TRIAL: NCT06464562
Title: LiveWell: An Adapted Dialectical Behavioral Therapy Skills Training Protocol for Patients Living With Metastatic Lung Cancer
Brief Title: LiveWell: Adapted DBT Skills Training for Metastatic Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00114867; 1K99CA286959 (NIH)
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Cancer Metastatic to Lung

STUDY DESIGN:
Intervention Model Description: Single arm for user testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LiveWell: Adapted Dialectical Behavioral Therapy Skills Training (Experimental): Participants randomized to LiveWell will receive the refined intervention protocol as informed by Aim 1 (K99). LiveWell is an 8-session protocol of Dialectical Behavioral Therapy Skills Training, adapted specifically for patients with metastatic lung cancer. Sessions are delivered one on one via telehealth, approximately weekly. Participants learn concrete, easy-to-use skills to: 1) tune into the present moment, and how they are thinking and feeling (mindfulness), understand emotions, how to change them, and how to experience more positive feelings (emotion regulation), tolerate distressing emotions and symptoms (e.g., fatigue, pain, dyspnea) and to accept reality as it is (distress tolerance), and tools to communicate wants and needs effectively with others (interpersonal effectiveness). The goal is to teach patients skills to live well, with metastatic cancer. All sessions follow a standardized structure that is customary in skills training and grounded in social cognitive theory.
  Interventions: Behavioral: LiveWell: Adapted Dialectical Behavioral Therapy Skills Training

INTERVENTIONS:
Behavioral: LiveWell: Adapted Dialectical Behavioral Therapy Skills Training — An adapted dialectical behavioral therapy skills training intervention

SUMMARY:
Patients are living longer with metastatic lung cancer (i.e., metavivors) due to therapeutic advances, but face significant challenges. Most metavivors will ultimately die of cancer and must navigate the duality of living while dying. Unsurprisingly, metavivors endorse high psychological distress (e.g., anxiety, depression, illness non-acceptance), high symptom burden (e.g., fatigue, dyspnea, pain), and poor quality of life. Psychosocial interventions can improve outcomes, but existing paradigms are not designed to help metavivors navigate the emotional turbulence of living with metastatic disease. Dialectical Behavioral Therapy (DBT) Skills Training is an evidence-based treatment that teaches patients transdiagnostic, easy-to-use skills to both accept things as they are (mindfulness, distress tolerance) and change things within their control (emotion regulation, interpersonal effectiveness) to better navigate life challenges. However, DBT Skills Training has rarely been applied in patients with chronic illness. The investigators adapted DBT Skills Training (e.g., intervention dose, delivery, content) for patients living with metastatic lung cancer to create LiveWell, an 8-session Skills Training protocol delivered one-on-one via videoconference. Building on preliminary data and aligned with the ORBIT model for behavioral intervention development, the first phase of this study (K99, Aim 1, 1 year) aims to iteratively refine LiveWell using 1) qualitative exit interview data from a proof-of-concept study, 2) an advisory board of interested parties, 3) the Dynamic Sustainability Framework from implementation science, and 4) user testing (n= up to 10). The K99 phase will produce a standardized protocol and procedures for the second, independent phase of the study (R00) which will be registered separately. If successful, LiveWell will improve metavivor quality of life and provide a promising psychosocial intervention paradigm for other metavivors and patients with chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with metastatic (AJCC stage IV) non-small cell lung cancer
* Undergoing lung cancer treatment with non-curative intent
* Endorse >=3 out of 10 on the NCCN distress thermometer over the past week
* At least 18 years of age
* Able to understand, speak, and read English, and 5) be able to provide informed consent

Exclusion Criteria:

* Reported or suspected cognitive impairment
* Presence of untreated serious mental illness (e.g., schizophrenia) indicated by the medical chart or treating oncologist
* Expected survival <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Somers, Principal Investigator — Professor in Psychiatry and Behavioral Sciences
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LiveWell: Adapted Dialectical Behavioral Therapy Skills Training: LiveWell is an 8-session protocol of Dialectical Behavioral Therapy Skills Training, adapted specifically for patients with metastatic lung cancer. Sessions are delivered one on one via telehealth, approximately weekly.
Period: Overall Study
Arm/Group | LiveWell: Adapted Dialectical Behavioral Therapy Skills Training
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LiveWell: Adapted Dialectical Behavioral Therapy Skills Training
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Usability as Measured by the Total Number of Participants Who Complete the Study Questionnaires
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | LiveWell: Adapted Dialectical Behavioral Therapy Skills Training
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | LiveWell: Adapted Dialectical Behavioral Therapy Skills Training
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT06464562/Prot_SAP_001.pdf
  • Informed Consent Form (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT06464562/ICF_000.pdf